CLINICAL TRIAL: NCT00659035
Title: Use of Driving Tests to Evaluate Patient Performance on Oral Opioids
Acronym: OpDrive
Status: Active, not recruiting | Type: Observational
Sponsor: Asokumar Buvanendran (Other)
Responsible Party: Sponsor-Investigator, Asokumar Buvanendran, Attending Physician, Associate Professor, Rush University Medical Center
Organization: Rush University Medical Center (Other)
Other Study IDs: ABuv111407
Record Dates: First submitted 2008-01-30; First posted 2008-04-16 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Chronic Pain
Keywords: driving; opioids; impairment; ability; patients; receiving; oral morphine; severe
MeSH Terms: conditions — Chronic Pain; Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- IT: Subjects receiving 1-10 mg/day of morphine or its equivalent doses of opioid medications through intrathecal route. Intrathecal medications are administered through a catheter in spinal cord
- Oral: Subjects receiving oral opioids (morphine, oxycodone, hydrocodone, methadone), but not also receiving anticonvulsants (gabapentin, pregabalin, topiramate), muscle relaxants, benzodiazepines, or diphenylhydramine for at least a week before testing; low dose antidepressants and/or NSAIDs are OK
- Oral + Anticonvulsant: Subjects receiving oral opioids (morphine, oxycodone, hydrocodone, methadone) and anticonvulsants (gabapentin, pregabalin, topiramate), but not also receiving muscle relaxants, benzodiazepines, or diphenylhydramine for at least a week before testing; low dose antidepressants and/or NSAIDs are OK
- Control -Pain: Subject not receiving opioid medications, anticonvulsants (gabapentin, pregabalin, topiramate), muscle relaxants, benzodiazepines, or diphenylhydramine for at least a week before testing; low dose antidepressants and/or NSAIDs are OK.
- Control -No Pain: Age-matched volunteers (NO PAIN) not receiving opioid medications, anticonvulsants (gabapentin, pregabalin, topiramate), muscle relaxants, benzodiazepines, or diphenylhydramine for at least a week before testing; low dose antidepressants and/or NSAIDs are OK.

SUMMARY:
Many patients seen at Pain Centers are advised not to drive if they are on long-term opioid medications. Although such advice is routinely given considering patients' safety, unnecessary restrictions to driving can cause inconvenience to the patients and delay their treatment. Such restrictions also pose social and legal questions to patients and physicians.

The investigators would like to test such patients' ability to drive under oral opioids using a driving simulator at the Pain Center. This simulator is like a video game with computer and a steering wheel to simulate real life driving. The driving simulator provides measure on several outcome measures, such as attention, reaction time, etc. allowing us to specifically address question pertaining to any cognitive or behavioral differences.

DETAILED DESCRIPTION:
Many patients seen at Pain Centers are advised not to drive if they are on long-term opioid medications. Although such advice is routinely given considering patients' safety, unnecessary restrictions to driving can cause inconvenience to the patients and delay their treatment. Such restrictions also pose social and legal questions to patients and physicians.

The investigators would like to test such patients' ability to drive under oral opioids using a driving simulator at the Pain Centre. This simulator is like a video game with computer and a steering wheel to simulate real life driving. The driving simulator provides measure on several outcome measures, such as attention, reaction time, etc. allowing us to specifically address question pertaining to any cognitive or behavioral differences.

A pilot phase, for feasibility, included 80 subjects. This phase will include a comparison with a random selection of 450 patients receiving one of the following 5 treatments:

Group 1 (IT): Subjects receiving 1-10 mg/day of morphine or its equivalent doses of opioid medications through intrathecal route. Intrathecal medications are administered through a catheter in spinal cord

Group 2 (Oral): Subjects receiving oral opioids (morphine, oxycodone, hydrocodone, methadone), but not also receiving anticonvulsants (gabapentin, pregabalin, topiramate), muscle relaxants, benzodiazepines, or diphenylhydramine for at least a week before testing; low dose antidepressants and/or NSAIDs are OK

Group 3 (Oral + Anticonvulsant): Subjects receiving oral opioids (morphine, oxycodone, hydrocodone, methadone) and anticonvulsants (gabapentin, pregabalin, topiramate), but not also receiving muscle relaxants, benzodiazepines, or diphenylhydramine for at least a week before testing; low dose antidepressants and/or NSAIDs are OK

Group 4 (Control -Pain) Subject not receiving opioid medications, anticonvulsants (gabapentin, pregabalin, topiramate), muscle relaxants, benzodiazepines, or diphenylhydramine for at least a week before testing; low dose antidepressants and/or NSAIDs are OK.

Group 5 (Control -No Pain) Age-matched volunteers (NO PAIN) not receiving opioid medications, anticonvulsants (gabapentin, pregabalin, topiramate), muscle relaxants, benzodiazepines, or diphenylhydramine for at least a week before testing; low dose antidepressants and/or NSAIDs are OK.

First group has 50 patients and the rest will have 100 patients each.

ELIGIBILITY:
Inclusion Criteria:

* Driving license

Exclusion Criteria:

* Any other drug or condition that would impair driving ability
* History of seizures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pain Clinic population
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2008-04 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Weaving, measured as standard deviation of lateral position. | 1 h

SECONDARY OUTCOMES:
Reaction time | 1 h

CONTACTS AND LOCATIONS:
Overall Officials: Asokumar Buvanendran, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States